CLINICAL TRIAL: NCT06308770
Title: Fatigue in Lupus Intervention Programmes (FLIP): A Randomised Controlled Trial Investigating the Effectiveness of Fatigue Management in Systemic Lupus Erythematosus
Brief Title: Fatigue in Lupus Intervention Programmes (FLIP)
Acronym: FLIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AC21137
Record Dates: First submitted 2024-02-23; First posted 2024-03-13 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Fatigue management
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Standard of Care; N-formylmethionylphenylalanine

STUDY DESIGN:
Intervention Model Description: The pilot study for the FLIP trial is a single centre three arm, randomised controlled trial (RCT) comparing the effectiveness of a virtual group fatigue management intervention with standard care in SLE participants. Participants will self-enrol via a secure database and then be randomised electronically to one of the three interventions;
  1. Standard care (SC) - Lupus UK and Versus Arthritis Booklets
  2. SC and 4 week Fatigue management Programme (FMP)
  3. SC and 7 week FMP Results will be measured by comparing Patient Reported Outcome measures (PROMs) submitted before and after the intervention and, at 6 and 12 months.
Who Masked: Outcomes Assessor
Masking Description: The statistician who analyses the results will be blind to the intervention to which the participant was randomised.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard care (Active Comparator): Participants will be provided with access to Versus Arthritis and Lupus UK fatigue booklets.
  Interventions: Behavioral: Standard Care
- Standard care and 4 week Fatigue Management Programme (FMP) (Active Comparator): Participants will be provided with access to Versus Arthritis and Lupus UK fatigue booklets and be randomised to a 4 week virtual FMP. They will attend live online group weekly sessions for 3 consecutive weeks followed by a review session at week 11.
  Interventions: Behavioral: Standard Care; Behavioral: 4 week FMP
- Standard care and 7 week Fatigue Management Programme (FMP) (Active Comparator): Participants will be provided with access to Versus Arthritis and Lupus UK fatigue booklets and be randomised to a 7 week virtual FMP. They will attend live online group weekly sessions for 6 consecutive weeks followed by a review session at week 14.
  Interventions: Behavioral: Standard Care; Behavioral: 7 week FMP

INTERVENTIONS:
Behavioral: Standard Care — Participants receive fatigue booklets from two charitable organisations providing information on fatigue, sleep, energy conservation, exercise and stress to help manage fatigue.
Behavioral: 4 week FMP — Participants attend 3 once weekly live online group interventions with a final intervention 8 weeks later.
  Arms: Standard care and 4 week Fatigue Management Programme (FMP)
Behavioral: 7 week FMP — Participants attend 6 once weekly live online group interventions with a final intervention 8 weeks later.
  Arms: Standard care and 7 week Fatigue Management Programme (FMP)

SUMMARY:
Systemic Lupus Erythematosus (SLE) is an autoimmune rheumatic disease. Patients report that fatigue has a significant impact on their quality of life but is often not discussed in healthcare settings. Fatigue is more prevalent in SLE than other Rheumatic diseases. Management across the NHS is very variable ranging from a booklet to one to one appointments or, less often, a group intervention. Previous studies in other Rheumatic diseases have shown that a group cognitive behavioural approach can be effective in helping patients manage their fatigue. The COVID-19 pandemic changed the way healthcare is delivered in the NHS . Healthcare professionals had to find alternate solutions e.g. Virtual appointments.

Our study aims to establish whether a virtual group Fatigue Management Programme and a fatigue booklet (Versus Arthritis and Lupus UK) is more effective at reducing the impact of fatigue in SLE participants than the fatigue booklet alone.

The investigators will also compare a shortened 4-week to the standard 7-week programme to lessen the time commitment for participants and potentially reduce waiting times.The investigators will measure the effectiveness of the interventions through the use of Patient Reported Outcome Measures (PROMs) at several intervals whilst the participant is enrolled in the study.The pilot study will run in a single site in Edinburgh. The investigators aim to find a manageable, cost effective solution for the NHS and patients to address this frequently unmet need.

DETAILED DESCRIPTION:
The FLIP study will recruit SLE patients to a single centre, three arm randomised controlled trial which will compare standard care ( fatigue booklets available in all Rheumatology departments in the UK or online ) with live online fatigue management groups for effectiveness at managing fatigue.

Lupus UK will advertise the study through their website, newsletter and social media. Participants can be identified and enrolled to the study in three ways:

1. The participant can be identified by any member of the Rheumatology department in NHS Lothian through participant routine Rheumatology appointment or local database. No patient records will be screened .
2. Participants can be identified through the Scottish Lupus Registry Database as they will have already consented to being contacted about research.
3. Participants can also self-enrol to the study through the link to the FLIP website from Lupus UK .

Posters, leaflets and LUPUS UK communications will have a link and QR code which will take interested participants to the patient information sheet to read about the study.They can contact the study team with any questions before proceeding to accessing the enrolment process in the REDCap secure server. The central study team or the participant themselves can confirm their eligibility by completing short screening questions.The study team can also help the patient with any questions regarding the online consent form if necessary. If the participant is eligible and wishes to proceed they will be asked to complete an online consent and be assigned a unique identification code number (UICN).

After the participant has consented online in REDCap and completed personal details/demographics and baseline PROMs questionnaires they will be randomised to either standard care, standard care plus 4 week programme or standard care plus 7 week programme. The ratio of randomisation will be 1.1.1 .

Participants will complete the same PROMS three more times after the baseline: on completion of the intervention, at 6 months and at 12 months.

The PROMs will be

1. Modified Fatigue Impact Score (MFIS)
2. SLE quality of life questionnaire (LupusQoL)
3. Pittsburgh Sleep quality Inventory ( PSQI)
4. Visual Analog scale of fatigue impact ( FI-VAS)
5. Participant health questionnaire -4 item (PHQ4)
6. Self -Efficacy for managing chronic disease 6 item scale (SEMCD-6)
7. Quick Systemic Lupus Activity Questionnaire (Q-SLAQ)

If a participant has access to a Systemic Lupus Erythematosus Disease Activity Index ( SLEDAI) score this may be included .

Participants will also be asked to complete a satisfaction questionnaire after the intervention completion.

The end of study is defined as the last data collection at 52 weeks from the last participant after group intervention or standard care whichever comes last.

The trial team will analyse the qualitative data from participants. A health economist will calculate the NHS utilisation / economic evaluation by mapping the LUPUSQoL to the Short Form 6 dimension (SF6D) to obtain quality adjusted life years (QALYs) .

A statistician will analyse the data from the PROMs with standard statistical software in R and report descriptive statistics such as means, medians, standard deviations and standard errors of the variables measured. Statistical significance will be measured for the aims of the study using unmatched and paired T- tests.

The primary outcome of our study, MFIS measurements, will be assessed using linear regression models including a random effect to account for grouping by centre. The investigators will assess whether the treatment outcome is maintained by analysing longitudinal data collected over 1 year using linear mixed-effect models with a suitable covariance structure. The secondary outcomes will be analysed in an analogous way. The investigators will also analyse how the secondary outcomes covary with the MFIS scores. The investigators will handle non-compliance by analysing the data according to intention-to-treat principles. In the unlikely event of unused data arising, the investigators will include these in suitable subgroup analyses. Spurious data will be followed up with patients and will only be excluded from the study as a measure of last resort. The investigators are not planning to carry out interim analyses nor to terminate the study early.

The results will be published in peer reviewed journals and by Lupus UK .

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed SLE Diagnosis
2. Be over 18 at time of consent
3. Report fatigue to be a chronic problem in the last 4 weeks with a VAS fatigue impact ≥ 6, based on a scale of 1 ( no fatigue impact on quality of life ) to 10 (severe impact of fatigue on quality of life).[20]
4. Agree to online consent, complete questionnaires and be randomised to standard care or group intervention programme via secure server (REDCap).
5. Not have taken part in a group fatigue or pain management programme in the past 5 years.
6. Have the ability to read and converse in English competently
7. Have access to a computer/Smartphone/Tablet for internet and audio/video access.
8. Be able to or willing to learn to use an NHS approved platform.
9. Be willing to provide a telephone, postal address and email address for communication related to the FLIP trial.

Exclusion Criteria:

1. They are unable to understand English sufficiently to attend a live online group programme. Facilitators and other group members will most likely only speak English.
2. They are unable to provide confirmation of eligibility, complete online informed consent or questionnaires
3. They are currently participating in an interventional trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Modified Fatigue Impact Score (MFIS) | 12 months
  A tool to measure the impact of fatigue including physical, cognitive, and psychosocial subscales. Scoring is 0-84, the higher the score the greater the impact of fatigue.

SECONDARY OUTCOMES:
Lupus quality of life questionnaire (LupusQoL) | 12 months
  A self-reported disease-specific health related quality of life questionnaire in adult Lupus. It consists of 34 items covering eight areas which include physical health, emotional health, body image, pain, planning, fatigue, intimate relationships, and burden to others. The questionnaire also has a 5-point Likert response format ranging from 0=all the time, 1=most of the time, 2=a good bit of the time, 3=occasionally, and 4=never. The higher the score the higher the reported quality of life.
Pittsburgh Sleep quality Inventory ( PSQI) | 12 months
  A self-rated questionnaire which measures sleep quality and sleep disturbances over a 1-month time period. There are 19 items which produce 7 "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The calculation of scores for these seven components produces one global score. If this score is greater than 5 it indicates poor sleep quality.
Visual Analog scale of fatigue impact (FI-VAS) | 12 months
  Designed by the researchers for this study, it is a 100mm horizontal line fastened by two statements representing extremes of a single range. The two statements in this VAS are Fatigue does /does not impact my life. A score of 100 mm indicates maximum impact of fatigue.
Participant Health Questionnaire (PHQ4) | 12 months
  A 4-item Likert response questionnaire using the first two items from the PHQ9 and GAD7 to briefly measure depression and anxiety. The brevity of the questionnaire was designed for clinical practice as a screening tool and is easier for participants who have fatigue and poor concentration. The maximum score is 12, a score of >8 indicates severe levels of distress.
Self-Efficacy for Managing Chronic Diseases 6-item Scale | 12 Months
  A 6 item scale on a visual analogue scale, ranging from 1 (not at all confident) to 10 (totally confident). The maximum score s 60.
Quick Systemic Lupus Erythematosus Activity Questionnaire (Q-SLAQ) | 12 months
  A shortened version of the Systemic Lupus Erythematosus Activity Questionnaire, a patient reported questionnaire of their Lupus related symptoms and disease activity. Maximum score is 37, the higher the score the higher the patient reported lupus activity.
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | 12 months
  A measure of disease activity in Lupus participants, calculated by a healthcare professional, based on symptoms experienced in the previous 10 days. The maximum score is 105, a score of 10 or above indicates high disease activity.

CONTACTS AND LOCATIONS:
Overall Officials: Helen Harris, BA MB BCh BAO, Principal Investigator — University of Edinburgh
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahn GE, Ramsey-Goldman R. Fatigue in systemic lupus erythematosus. Int J Clin Rheumtol. 2012 Apr 1;7(2):217-227. doi: 10.2217/IJR.12.4. PMID 22737181
- [Background] Azizoddin DR, Gandhi N, Weinberg S, Sengupta M, Nicassio PM, Jolly M. Fatigue in systemic lupus: the role of disease activity and its correlates. Lupus. 2019 Feb;28(2):163-173. doi: 10.1177/0961203318817826. Epub 2018 Dec 22. PMID 30580659
- [Background] Arnaud L, Gavand PE, Voll R, Schwarting A, Maurier F, Blaison G, Magy-Bertrand N, Pennaforte JL, Peter HH, Kieffer P, Bonnotte B, Poindron V, Fiehn C, Lorenz H, Amoura Z, Sibilia J, Martin T. Predictors of fatigue and severe fatigue in a large international cohort of patients with systemic lupus erythematosus and a systematic review of the literature. Rheumatology (Oxford). 2019 Jun 1;58(6):987-996. doi: 10.1093/rheumatology/key398. PMID 30597077
- [Background] Wang B, Gladman DD, Urowitz MB. Fatigue in lupus is not correlated with disease activity. J Rheumatol. 1998 May;25(5):892-5. PMID 9598886
- [Background] Nikiphorou E, Santos EJF, Marques A, Bohm P, Bijlsma JW, Daien CI, Esbensen BA, Ferreira RJO, Fragoulis GE, Holmes P, McBain H, Metsios GS, Moe RH, Stamm TA, de Thurah A, Zabalan C, Carmona L, Bosworth A. 2021 EULAR recommendations for the implementation of self-management strategies in patients with inflammatory arthritis. Ann Rheum Dis. 2021 Oct;80(10):1278-1285. doi: 10.1136/annrheumdis-2021-220249. Epub 2021 May 7. PMID 33962964
- [Background] Hewlett S, Almeida C, Ambler N, Blair PS, Choy E, Dures E, Hammond A, Hollingworth W, Kadir B, Kirwan J, Plummer Z, Rooke C, Thorn J, Turner N, Pollock J. Group cognitive-behavioural programme to reduce the impact of rheumatoid arthritis fatigue: the RAFT RCT with economic and qualitative evaluations. Health Technol Assess. 2019 Oct;23(57):1-130. doi: 10.3310/hta23570. PMID 31601357
- [Background] Hewlett S, Almeida C, Ambler N, Blair PS, Choy EH, Dures E, Hammond A, Hollingworth W, Kadir B, Kirwan JR, Plummer Z, Rooke C, Thorn J, Turner N, Pollock J; RAFT Study Group. Reducing arthritis fatigue impact: two-year randomised controlled trial of cognitive behavioural approaches by rheumatology teams (RAFT). Ann Rheum Dis. 2019 Apr;78(4):465-472. doi: 10.1136/annrheumdis-2018-214469. Epub 2019 Feb 6. PMID 30793700
- [Background] Martin KR, Bachmair EM, Aucott L, Dures E, Emsley R, Gray SR, Hewlett S, Kumar V, Lovell K, Macfarlane GJ, MacLennan G, McNamee P, Norrie J, Paul L, Ralston S, Siebert S, Wearden A, White PD, Basu N. Protocol for a multicentre randomised controlled parallel-group trial to compare the effectiveness of remotely delivered cognitive-behavioural and graded exercise interventions with usual care alone to lessen the impact of fatigue in inflammatory rheumatic diseases (LIFT). BMJ Open. 2019 Jan 30;9(1):e026793. doi: 10.1136/bmjopen-2018-026793. PMID 30705244
- [Background] Bachmair EM, Martin K, Aucott L, Dhaun N, Dures E, Emsley R, Gray SR, Kidd E, Kumar V, Lovell K, MacLennan G, McNamee P, Norrie J, Paul L, Packham J, Ralston SH, Siebert S, Wearden A, Macfarlane G, Basu N; LIFT study group. Remotely delivered cognitive behavioural and personalised exercise interventions for fatigue severity and impact in inflammatory rheumatic diseases (LIFT): a multicentre, randomised, controlled, open-label, parallel-group trial. Lancet Rheumatol. 2022 Jun 27;4(8):e534-e545. doi: 10.1016/S2665-9913(22)00156-4. eCollection 2022 Aug. PMID 36388001
- [Background] O'Riordan R, Doran M, Connolly D. Fatigue and Activity Management Education for Individuals with Systemic Lupus Erythematosus. Occup Ther Int. 2017 Jan 11;2017:4530104. doi: 10.1155/2017/4530104. eCollection 2017. PMID 29097965
- [Background] Carandang K, Poole J, Connolly D. Fatigue and activity management education for individuals with systemic sclerosis: Adaptation and feasibility study of an intervention for a rare disease. Musculoskeletal Care. 2022 Sep;20(3):593-604. doi: 10.1002/msc.1617. Epub 2022 Feb 6. PMID 35124888
- [Background] Fangtham M, Kasturi S, Bannuru RR, Nash JL, Wang C. Non-pharmacologic therapies for systemic lupus erythematosus. Lupus. 2019 May;28(6):703-712. doi: 10.1177/0961203319841435. Epub 2019 Apr 8. PMID 30961418
- [Background] Overman CL, Kool MB, Da Silva JA, Geenen R. The prevalence of severe fatigue in rheumatic diseases: an international study. Clin Rheumatol. 2016 Feb;35(2):409-15. doi: 10.1007/s10067-015-3035-6. Epub 2015 Aug 15. PMID 26272057
- [Background] Meacock R, Harrison M, McElhone K, Abbott J, Haque S, Bruce I, Teh LS. Mapping the disease-specific LupusQoL to the SF-6D. Qual Life Res. 2015 Jul;24(7):1749-58. doi: 10.1007/s11136-014-0892-4. Epub 2014 Dec 16. PMID 25510215
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Harris PA, Taylor R, Minor BL, Elliott V, Fernandez M, O'Neal L, McLeod L, Delacqua G, Delacqua F, Kirby J, Duda SN; REDCap Consortium. The REDCap consortium: Building an international community of software platform partners. J Biomed Inform. 2019 Jul;95:103208. doi: 10.1016/j.jbi.2019.103208. Epub 2019 May 9. PMID 31078660
- [Background] Larson RD. Psychometric properties of the modified fatigue impact scale. Int J MS Care. 2013 Spring;15(1):15-20. doi: 10.7224/1537-2073.2012-019. PMID 24453758
- [Background] Yazdany J. Health-related quality of life measurement in adult systemic lupus erythematosus: Lupus Quality of Life (LupusQoL), Systemic Lupus Erythematosus-Specific Quality of Life Questionnaire (SLEQOL), and Systemic Lupus Erythematosus Quality of Life Questionnaire (L-QoL). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11(0 11):S413-9. doi: 10.1002/acr.20636. No abstract available. PMID 22588761
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Hewlett S, Dures E, Almeida C. Measures of fatigue: Bristol Rheumatoid Arthritis Fatigue Multi-Dimensional Questionnaire (BRAF MDQ), Bristol Rheumatoid Arthritis Fatigue Numerical Rating Scales (BRAF NRS) for severity, effect, and coping, Chalder Fatigue Questionnaire (CFQ), Checklist Individual Strength (CIS20R and CIS8R), Fatigue Severity Scale (FSS), Functional Assessment Chronic Illness Therapy (Fatigue) (FACIT-F), Multi-Dimensional Assessment of Fatigue (MAF), Multi-Dimensional Fatigue Inventory (MFI), Pediatric Quality Of Life (PedsQL) Multi-Dimensional Fatigue Scale, Profile of Fatigue (ProF), Short Form 36 Vitality Subscale (SF-36 VT), and Visual Analog Scales (VAS). Arthritis Care Res (Hoboken). 2011 Nov;63 Suppl 11:S263-86. doi: 10.1002/acr.20579. No abstract available. PMID 22588750
- [Background] Kroenke K, Spitzer RL, Williams JB, Lowe B. An ultra-brief screening scale for anxiety and depression: the PHQ-4. Psychosomatics. 2009 Nov-Dec;50(6):613-21. doi: 10.1176/appi.psy.50.6.613. PMID 19996233
- [Background] Lorig KR, Sobel DS, Ritter PL, Laurent D, Hobbs M. Effect of a self-management program on patients with chronic disease. Eff Clin Pract. 2001 Nov-Dec;4(6):256-62. PMID 11769298
- [Background] Svenungsson E, Gunnarsson I, Illescas-Backelin V, Trysberg E, Jonsen A, Leonard D, Sjowall C, Pettersson S. Quick Systemic Lupus Activity Questionnaire (Q-SLAQ): a simplified version of SLAQ for patient-reported disease activity. Lupus Sci Med. 2021 May;8(1):e000471. doi: 10.1136/lupus-2020-000471. PMID 33972457
- [Background] Cleanthous S, Tyagi M, Isenberg DA, Newman SP. What do we know about self-reported fatigue in systemic lupus erythematosus? Lupus. 2012 Apr;21(5):465-76. doi: 10.1177/0961203312436863. Epub 2012 Feb 16. PMID 22345120
- [Background] Hewlett S, Ambler N, Almeida C, Blair PS, Choy E, Dures E, Hammond A, Hollingworth W, Kirwan J, Plummer Z, Rooke C, Thorn J, Tomkinson K, Pollock J; RAFT Study Team. Protocol for a randomised controlled trial for Reducing Arthritis Fatigue by clinical Teams (RAFT) using cognitive-behavioural approaches. BMJ Open. 2015 Aug 6;5(8):e009061. doi: 10.1136/bmjopen-2015-009061. PMID 26251413
- [Background] Cervilla O, Miro E, Martinez MP, Sanchez AI, Sabio JM, Prados G. Sleep quality and clinical and psychological manifestations in women with mild systemic lupus erythematosus activity compared to women with fibromyalgia: A preliminary study. Mod Rheumatol. 2020 Nov;30(6):1016-1024. doi: 10.1080/14397595.2019.1679973. Epub 2019 Nov 14. PMID 31599659
- [Background] Xerfan EMS, Andersen ML, Tomimori J, Tufik S, Facina AS. The role of sleep in the activity of lupus erythematosus: an overview of this possible relationship. Rheumatology (Oxford). 2021 Feb 1;60(2):483-486. doi: 10.1093/rheumatology/keaa744. No abstract available. PMID 33241379
- [Background] Fenn, K. and M. Byrne, The key principles of cognitive behavioural therapy. InnovAiT: Education and inspiration for general practice, 2013. 6(9): p. 579-585.
- [Background] Lee, D.R., Teaching the World to Sleep. 2018.
- [Result] Dobson, J., et al., POS1496-HPR HARD TIMES: ADAPTING A FATIGUE MANAGEMENT PROGRAMME IN A PANDEMIC. Annals of the Rheumatic Diseases, 2022. 81(Suppl 1): p. 1093-1093.
- See also: prevalence of severe fatigue in Lupus — http://www.webmd.com/lupus/lupus-fatigue
- See also: prevalence of SLE in the UK — http://www.cprd.com/protocol/epidemiology-systemic-lupus-erythematosus-sle-and-lupus-nephritis-ln-england-retrospective
- See also: Versus Arthritis booklet on fatigue — http://www.versusarthritis.org/media/23151/fatigue-and-arthritis-information-booklet.pdf